CLINICAL TRIAL: NCT07103772
Title: Effect of Consuming a Nutraceutical Composition Based on Pineapple and Natural Extracts on Signs and Symptoms in Adult Patients With Irritable Bowel Syndrome
Brief Title: Effect of Consuming a Nutraceutical Composition on Signs and Symptoms in Adult Patients With Irritable Bowel Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Adbel Zaid Martínez Baez, Sciences' Doctor, Universidad Autonoma de Nuevo Leon
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-FaSPyN-AG-06
Record Dates: First submitted 2025-02-10; First posted 2025-08-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome With Constipation; Irritable Bowel Syndrome Mixed
Keywords: Síndrome del intestino irritable; Piña; Nuez; Guayaba; Intestino; Suplemento dietético; Antiinflamación; Efecto digestivo; Digestión
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison between two groups: nutraceutical and placebo treatment.
Who Masked: Participant, Investigator
Masking Description: For the purposes of the study, it was decided to use a double-blind method, where neither the investigator nor the patient knows which treatment is the nutraceutical and which is the placebo. To achieve this, the team was responsible for mixing the treatment packages to allow for proper distribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ananá´s Nutraceutical Goup (Experimental): 47 personas recibirán el tratamiento de 14 días con el suplemento nutracéutico.
  Interventions: Dietary Supplement: Ananá
- Ananá´s Placebo Group (Placebo Comparator): 47 people will recieve the 14 day treatment with the placebo supplement.
  Interventions: Dietary Supplement: Ananá

INTERVENTIONS:
Dietary Supplement: Ananá — The supplement consists of a box containing 14 sachets of the product for 14 days of treatment. Patients should preferably consume the supplement in the morning.
  The "Ananá's Nutraceutical Group" will receive the real supplement for consumption over 14 days, while the "Ananá's Placebo Group" will receive a placebo supplement for comparison at the end of the trial.

SUMMARY:
Irritable bowel syndrome is characterized by the presence of chronic, recurrent abdominal pain, alterations in bowel habits, and abdominal distension. The medical diagnosis is made using the Rome IV criteria. There are three IBS phenotypes: diarrhea-predominant, constipation-predominant, and mixed.

DETAILED DESCRIPTION:
A sample of 100 people will be supplemented, with 50 participants consuming the nutraceutical gel and the remaining 50 receiving a placebo supplement. The supplementation period lasts 14 days, during which severity questionnaires and the Bristol Stool Scale will be administered on Day 0, Day 7, and Day 14. Additionally, to assess biomarkers, biochemical tests for PCR, calprotectin, and fecal lactoferrin will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years old.
* Be an employee or beneficiary of UANL.
* Have gastrointestinal alterations (diarrhea, constipation, etc.) that suggest the presence of irritable bowel syndrome.
* Not be under any medical treatment.

Exclusion Criteria:

* Being under medical treatment.
* Not having gastrointestinal alterations much as diarrhea, constipation, etc.
* being under 18 years old.
* Not being an employee or beneficiary of UANL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female.
Enrollment: 94 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Effect of the Consumption of a Nutraceutical Composition on Signs and Symptoms in Adult Patients with Irritable Bowel Syndrome. | 1 year
  A sample of 100 people will be supplemented, with 50 participants consuming the nutraceutical gel and the remaining 50 receiving a placebo supplement. The supplementation period lasts 14 days, during which severity questionnaires and the Bristol Stool Scale will be administered on Day 0, Day 7, and Day 14. Additionally, to assess biomarkers, biochemical tests for PCR, calprotectin, and fecal lactoferrin will be conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
The personal data, including biochemical data of the participants, will not be shared for use in other clinical trials or for additional research purposes.

REFERENCES:
- [Background] Menees SB, Powell C, Kurlander J, Goel A, Chey WD. A meta-analysis of the utility of C-reactive protein, erythrocyte sedimentation rate, fecal calprotectin, and fecal lactoferrin to exclude inflammatory bowel disease in adults with IBS. Am J Gastroenterol. 2015 Mar;110(3):444-54. doi: 10.1038/ajg.2015.6. Epub 2015 Mar 3. PMID 25732419
- [Background] Kansakar U, Trimarco V, Manzi MV, Cervi E, Mone P, Santulli G. Exploring the Therapeutic Potential of Bromelain: Applications, Benefits, and Mechanisms. Nutrients. 2024 Jun 28;16(13):2060. doi: 10.3390/nu16132060. PMID 38999808
- [Background] Liu YM, Lin IJ, Huang CW, Chien RC, Mau CZ, Mau JL. Effect of Ethanolic Extracts from Taiwanofungus camphoratus and T. salmoneus (Agaricomycetes) Mycelia on Osteoporosis Recovery. Int J Med Mushrooms. 2020;22(3):277-287. doi: 10.1615/IntJMedMushrooms.2020033983. PMID 32479022
- [Background] Dai K, Agarwal N, Rodriguez-Palacios A, Basson AR. Regulation of Intestinal Inflammation by Walnut-Derived Bioactive Compounds. Nutrients. 2024 Aug 10;16(16):2643. doi: 10.3390/nu16162643. PMID 39203780
- [Background] Borrelli F, Capasso R, Severino B, Fiorino F, Aviello G, De Rosa G, Mazzella M, Romano B, Capasso F, Fasolino I, Izzo AA. Inhibitory effects of bromelain, a cysteine protease derived from pineapple stem (Ananas comosus), on intestinal motility in mice. Neurogastroenterol Motil. 2011 Aug;23(8):745-e331. doi: 10.1111/j.1365-2982.2011.01735.x. Epub 2011 Jun 21. PMID 21689210
- [Background] Ballou S, Singh P, Nee J, Rangan V, Iturrino J, Geeganage G, Lowe B, Bangdiwala SI, Palsson OS, Sperber AD, Lembo A, Lehmann M. Prevalence and Associated Factors of Bloating: Results From the Rome Foundation Global Epidemiology Study. Gastroenterology. 2023 Sep;165(3):647-655.e4. doi: 10.1053/j.gastro.2023.05.049. Epub 2023 Jun 13. PMID 37315866
- [Background] Bakare AO, Owoyele BV. Bromelain reduced pro-inflammatory mediators as a common pathway that mediate antinociceptive and anti-anxiety effects in sciatic nerve ligated Wistar rats. Sci Rep. 2021 Jan 11;11(1):289. doi: 10.1038/s41598-020-79421-9. PMID 33432004
- [Background] Oka P, Parr H, Barberio B, Black CJ, Savarino EV, Ford AC. Global prevalence of irritable bowel syndrome according to Rome III or IV criteria: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):908-917. doi: 10.1016/S2468-1253(20)30217-X. Epub 2020 Jul 20. PMID 32702295